CLINICAL TRIAL: NCT03486470
Title: Comparison of Two Radial Artery Segments Related to "Old-Fashioned" Radial and New Snuff Box Vessel Approach. Ultrasound Study of Both Arms
Brief Title: Comparison of Two Radial Artery Segments Related to "Old-Fashioned" Radial and New Snuff Box Vessel Approach by US
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Stephan Cherkezov Hospital (Other)
Responsible Party: Principal Investigator, Dr. Valentin Krastev, Head of CathLab, Dr. Stephan Cherkezov Hospital
Other Study IDs: MBVT-0218-1
Record Dates: First submitted 2018-02-28; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound examination of radial arteries — Measuring the diameter and the depth of two radial segments on both arms

SUMMARY:
The purpose of this study is to determine if there is a difference in the size and the depth of the radial artery at the access points for established radial and new distal radial approach for the arteries of both arms

DETAILED DESCRIPTION:
Radial approach for coronary and peripheral procedures is now well established due to both patient and operator preference and carries a lower risk of bleeding and mortality. The most lasting consequence of transradial procedures remains radial artery occlusion, which is mainly influenced by the artery diameter and the size of the sheath. As a new, more distal approach looms on the horizon, it is plausible to determine factors that could impact its feasibility. Since the success rate for artery cannulation depends to a great extent on the size and the depth of the artery, the current study examines both parameters, as well as whether they are influenced by variables such as sex, body mass index, handedness, or comorbidities i.e. diabetes mellitus and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old admitted to the Cardiology Department

Exclusion Criteria:

* Previous transradial procedures
* Arm AV fistula for dialysis access
* History of upper limb peripheral arterial disease
* Hemiparesis
* Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Cardilogy Department
Sampling Method: Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2018-08-15 (Estimated); Study Completion 2018-08-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of ultrasound derived diameters of radial artery measured at sites related to two different transradial arterial approaches for catheterization | 1 day
  Measuring diameters of the radial artery at the access points for well established radial and new distal radial approach and finding or not a significant difference could have some implications for choosing the access radial site. At the end of a routine echocardiographic evaluation, four short axis measurements (one proximal and one distal on each arm) of the radial artery diameters will be done with a vascular probe.

SECONDARY OUTCOMES:
Comparison of ultrasound derived depth of radial artery measured at sites related to two different transradial arterial approaches for catheterization | 1 day
  At the end of a routine echocardiographic evaluation, four measurements (one proximal and one distal on each arm) of the radial artery depth will be done with a vascular probe in a neutral position of the hand.
Impact of sex, BMI, hand-dominance or comorbidities on the size and the depth of the arterial segments | 1 day
  To determine if sex, BMI, hand-dominance and widespread comorbidities (hypertension and diabetes mellitus) influence the size and the depth of the radial artery

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Krastev, MD, Principal Investigator — Dr. Stephan Cherkezov Hospital; Haralamby Benov, MD, Principal Investigator — Dr. Stephan Cherkezov Hospital

IPD SHARING:
Plan to Share IPD: Undecided